CLINICAL TRIAL: NCT02345278
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine Tolerability and Safety of Different Dosages of SUBLIVAC FIX Mite Mixture in Patients With Allergic Rhinitis / Rhinoconjunctivitis Caused by House Dust Mites
Brief Title: SUBLIVAC FIX Mite Mixture Dose Tolerability Study
Acronym: DTS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HAL Allergy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SM/0044
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: House Dust Mite Allergy
Keywords: Immunotherapy; Allergic rhinitis/rhinoconjunctivitis
MeSH Terms: conditions — Dust Mite Allergy; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): once daily sublingual administration for 1 month
  Interventions: Other: Placebo
- SUBLIVAC FIX Mite mixture 10,000 AU/mL (Active Comparator): once daily sublingual administration for 1 month
  Interventions: Drug: SUBLIVAC FIX Mite mixture
- SUBLIVAC FIX Mite mixture 25,000 AU/mL (Active Comparator): once daily sublingual administration for 1 month
  Interventions: Drug: SUBLIVAC FIX Mite mixture
- SUBLIVAC FIX Mite mixture 50,000 AU/mL (Active Comparator): once daily sublingual administration for 1 month
  Interventions: Drug: SUBLIVAC FIX Mite mixture
- SUBLIVAC FIX Mite mixture 100,000 AU/mL (Active Comparator): once daily sublingual administration for 1 month
  Interventions: Drug: SUBLIVAC FIX Mite mixture

INTERVENTIONS:
Drug: SUBLIVAC FIX Mite mixture — Study medication will be taken sublingually once a day. Patients will start with one drop and increase the dose by one drop each consecutive day until the maintenance dose (5 drops/day) is reached. Drops should be kept under the tongue for 2-3 minutes before swallowing. After reaching the maintenance dose patients will be treated up to 1 month.
  Arms: SUBLIVAC FIX Mite mixture 10,000 AU/mL; SUBLIVAC FIX Mite mixture 100,000 AU/mL; SUBLIVAC FIX Mite mixture 25,000 AU/mL; SUBLIVAC FIX Mite mixture 50,000 AU/mL
Other: Placebo — Study medication will be taken sublingually once a day. Patients will start with one drop and increase the dose by one drop each consecutive day until the maintenance dose (5 drops/day) is reached. Drops should be kept under the tongue for 2-3 minutes before swallowing. After reaching the maintenance dose patients will be treated up to 1 month.
  Arms: Placebo

SUMMARY:
Allergic rhinitis/rhinoconjunctivitis is a symptomatic disorder of the nose induced by an immunoglobulin E (IgE) mediated inflammatory response. Treatment may involve pharmacotherapy and specific immunotherapy (IT). IT represents the only treatment that might alter the natural course of the disease. The amount of administered allergen is crucial for both efficacy and safety of specific IT. SUBLIVAC FIX Mite mixture is a preparation for sublingual IT (SLIT) and is indicated for the treatment of allergic disorders such as allergic rhinitis and rhinoconjunctivitis, caused by sensitisation to house dust mite (HDM) allergens.

According to the European Medicines Agency Guideline on the clinical development of products for specific IT for the treatment of allergic diseases, products should be tested at different dosages to provide preliminary data on safety and tolerability with regard to the maximum tolerated dose and suitable dose escalation scheme. This trial is designed to investigate the tolerability and safety of different dosages of SUBLIVAC FIX Mite mixture.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male or female patients, age ≥ 18 ≤ 60 years
3. Patients with allergic rhinitis or rhinoconjunctivitis induced by HDM for at least 1 year, with or without concomitant at least partly controlled asthma
4. Patients with a history of concomitant asthma should have a FEV1 > 70% (of predicted value) at inclusion. Patients without a history of asthma should have a FEV1 > 70% or a PEF > 80% (of predicted value)
5. Positive SPT to HDM D. pter or D. far (mean wheal diameter ≥ 3 mm compared to negative control; negative control should be negative; histamine control should be positive (mean wheal diameter ≥ 3 mm) at screening
6. Allergen specific serum IgE (ssIgE) level in serum for HDM D. pter or D. far (> 0.7 U/ml), assessed at screening

Exclusion Criteria:

1. Patients with concomitant sensitization i.e. positive SPT (mean wheal diameter ≥ 3 mm compared to negative control; negative control should be negative; histamine control should be positive (mean wheal diameter ≥ 3 mm) who are expected to have clinically relevant symptoms during the treatment period
2. Patients sensitized and symptomatic to pets who are regularly exposed to pets
3. Completed allergen-specific immunotherapy (SCIT or SLIT) with HDM within the last 5 years
4. Completed unsuccessful allergen-specific immunotherapy (SCIT or SLIT) within the last 5 years
5. Allergen-specific immunotherapy (SCIT or SLIT) with other allergens than HDM during the study period
6. Any other vaccination one week before start of treatment and during the up-dosing phase
7. Any anti-IgE therapy within the last 6 months prior to inclusion and during study
8. Active inflammatory disease in the mouth (e.g periodontitis, oral mucosal lichen planus)
9. Known hypersensitivity to any of the excipients (i.e. Disodium phosphate dihydrate, Sodium dihydrogen phosphate dihydrate, Aminocaproic acid, Glycerol, Peppermint oil, Caramel Colorant) of SLIT solution
10. Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
11. Active malignancies or any malignant disease in the last 5 years
12. A chronic or acute disease that in the opinion of the investigator might place the patient at an additional risk, including but not limited to the following: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine disorders, clinically significant renal or hepatic diseases, or haematological disorders
13. Diseases with a contra-indication for the use of adrenaline (e.g. hyperthyroidism, glaucoma)
14. Use of systemic corticosteroids 4 weeks before start treatment
15. Treatment with systemic or local beta-blockers
16. Clinically significant chronic sinusitis or ocular infection
17. Participation in a clinical study with a new investigational drug within the last 3 months or a biological within the last 6 months prior to the study or during the study
18. Pregnancy, lactation or inadequate contraceptive measures (acceptable forms of birth control include Intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections) or condom combined with a diaphragm including spermicidal cream). Also acceptable for women is surgical sterilization (removal of the uterus or ovaries or tubal ligation ("tied tubes")), if they are postmenopausal (12 consecutive months without a period) for at least 2 years, or having no sexual relationship with a man.
19. Alcohol, drug, or medication abuse within the past year and during the study
20. Any lack of co-operation or compliance
21. Severe psychiatric, psychological, or neurological disorders
22. Patients who are employees of the department or study site; 1st grade relatives, partners of the investigator, or patients who are dependent on the sponsor
23. Any physical or mental condition that precludes administration of allergen-specific immunotherapy, compliance or participation in a trial
24. Patients who are placed in an institution due to governmental or judicial directive

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SUBLIVAC FIX Mite mixture (assessed by number and severity of local and systemic reactions) | 1 month treatment
  Safety and tolerability of different dosages of SUBLIVAC FIX Mite mixture compared to placebo assessed by number and severity of local and systemic reactions.

SECONDARY OUTCOMES:
Adverse Events | 1 month treatment
  Safety of different dosages of SUBLIVAC FIX Mite mixture compared to placebo assessed by number and severity of Adverse Events
Clinical and laboratory parameters (Safety of different dosages of SUBLIVAC FIX Mite mixture) | 1 month treatment
  Safety of different dosages of SUBLIVAC FIX Mite mixture compared to placebo assessed by clinical and laboratory parameters
Changes in immunoglobulin levels ((IgE, IgG, IgG4) | 1 month
  Changes in serum specific immunoglobulin levels (IgE, IgG, IgG4) after 1 month of treatment with different dosages of SUBLIVAC FIX Mite mixture compared to placebo
Proportion of patients reaching maintenance dose within 10 days | 10 days
  Proportions of patients in the different treatment groups reaching maintenance dose within 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof.Dr.med., Study Chair — Allergie-Centrum-Charité
Locations (10):
- Germany (10):
  - Charite Universitatsmedizin Berlin, Allergiezentrum, Berlin
  - Praxis Dr.med.Elke Hippke, Berlin
  - HNO-Heilkunde Praxis, Chemnitz
  - HNO und Allergologie Praxis, Dresden
  - HNO-Praxis Dr. Uta Thieme, Duisburg
  - Universitatsklinikum Dusseldorf, Department Dermatology, Düsseldorf
  - HNO Praxis Gottingen, Göttingen
  - HNO Praxis am Neckar, Heidelberg
  - HNO Gemeinschaftspraxis, Heidelberg
  - Dr.med. Ulrich Neumann Praxis, Wolmirstedt